CLINICAL TRIAL: NCT02085317
Title: Observation of Microcirculation Impairment in Patients With Lepromatous Leprosy Using Orthogonal Polarization Spectral (OPS) Imaging and Laser Doppler Iontophoresis
Brief Title: Microcirculatory Impairment in Patients With Leprosy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Curt Treu (Other)
Responsible Party: Sponsor-Investigator, Curt Treu, Prof. Curt Treu, Rio de Janeiro State University
Organization: Rio de Janeiro State University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Biovasc-1
Record Dates: First submitted 2014-03-02; First posted 2014-03-12 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Lepromatous Leprosy
Keywords: Microcirculation; Leprosy; Nervous system; Orthogonal polarization spectral (OPS) imaging; Laser Doppler flowmetry; Iontophoresis.
MeSH Terms: conditions — Leprosy, Lepromatous; Leprosy; Neurologic Manifestations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lepromatous Patients (Other): Composed of patients with lepromatous Leprosy acetylcholine Iontophoresis sodium nitroprusside Iontophoresis
  Interventions: Drug: acetylcholine Iontophoresis; Drug: sodium nitroprusside Iontophoresis
- Healthy Patients (Other): Composed of patients without any disease acetylcholine Iontophoresis sodium nitroprusside Iontophoresis
  Interventions: Drug: acetylcholine Iontophoresis; Drug: sodium nitroprusside Iontophoresis

INTERVENTIONS:
Drug: acetylcholine Iontophoresis — Using a protocol similar to the one developed by Rossi and co-workers (Rossi et al., 2008), ACh (Acetylcholine - Sigma-Aldrich, St. Louis, USA) was delivered by 9 iontophoretic pulses of 0.1 mA for 20 s with 60 s interval between pulses using a drug delivery electrode filled with 0.1 ml of 1% ACh solution, attached to the dorsal aspect of the second left finger by a double-sided adhesive disc.
Drug: sodium nitroprusside Iontophoresis — After Ach, SNP (Nipride® 10mg/ml - Biolab, São Paulo, Brazil) was delivered by 7 iontophoretic pulses of 0.2 mA for 20 s with 180 s interval between pulses using another drug delivery electrode filled with 0.1 ml of 1% SNP solution, attached to the dorsal aspect of the third left finger. In both situations, an indifferent electrode was attached on the dorsal aspect of the left hand. Endothelial-dependent and independent skin vasodilator response to each iontophoresis pulse was measured in PUs, as mean value during each interval from one pulse to the following one.

SUMMARY:
In this study the investigators have aimed to evaluate morphology and reactivity of cutaneous microcirculation in patients with lepromatous leprosy. Ten patients, without any other comorbidity were compared to ten controls without leprosy or any other comorbidity, using the Cytoscan® [orthogonal polarization spectral (OPS) imaging], Fourier analysis of laser Doppler signal to evaluate vasomotion (rhythmic spontaneous oscillation of arteriolar diameter) and laser Doppler flowmetry associated to iontophoresis of vasoactive substances (acetylcholine and sodium nitroprusside).

DETAILED DESCRIPTION:
Evaluation with OPS:

After acclimatization, the microcirculation of patients and controls was assessed by OPS in three different points, according to criteria recommended by De Backer(De Backer et al., 2007). Images were recorded for 10 seconds at each point and evaluated afterwards using Cap-Image v7.2software.

Evaluation with laser-Doppler flowmetry (LDF):

Skin blood perfusion was measured in conventional perfusion units (PU) by means of a LDF apparatus (Periflux PF4, Perimed, Stockholm, Sweden), equipped with a non-heated probe (PF408), fixed to the medial surface of the right forearm. Laser characteristics were: 780 nm wavelength, 10-19 kHz bandwidth, 0.1 s time constant and 32 Hz sampling frequency. Skin blood perfusion was expressed in conventional perfusion units (PU: 1 PU=10 mV) and LD signal was recorded continuously by an interfaced computer (Sony VaioVGN-CR160A) equipped with Perisoft dedicated software. Exams were performed in two steps:

First, to register vasomotion, a probe (Probe 481-1: Single Iontophoresis Probe - Perimed, Stockholm, Sweden) was placed, after the skin was cleaned with a wipe of 70° alcohol and left to air dry, in the dorsal face of the distal phalanx of the 2nd finger. The probes were positioned at least 10 cm apart, avoiding superficial veins and broken skin areas. This probe may be used for both vasomotion and iontophoresis. Basal blood perfusion was continuously recorded during 20 min. Skin temperature was continuously measured.

To avoid residual effects of previously used drugs, the probe position for combined iontophoresis and LDF recordings were placed in untreated fingers [2nd for acetylcholine (Ach) and 3nd for sodium nitroprusside (SNP)] after each measurement .

Using a protocol similar to the one developed by Rossi and co-workers (Rossi et al., 2008), ACh (Acetylcholine - Sigma-Aldrich, St. Louis, USA) was delivered by 9 iontophoretic pulses of 0.1 mA for 20 s with 60 s interval between pulses using a drug delivery electrode filled with 0.1 ml of 1% ACh solution, attached to the dorsal aspect of the second left finger by a double-sided adhesive disc. After Ach, SNP (Nipride® 10mg/ml - Biolab, São Paulo, Brazil) was delivered by 7 iontophoretic pulses of 0.2 mA for 20 s with 180 s interval between pulses using another drug delivery electrode filled with 0.1 ml of 1% SNP solution, attached to the dorsal aspect of the third left finger. In both situations, an indifferent electrode was attached on the dorsal aspect of the left hand. Endothelial-dependent and independent skin vasodilator response to each iontophoresis pulse was measured in PUs, as mean value during each interval from one pulse to the following one.

ELIGIBILITY:
Inclusion Criteria:

* male patients with only lepromatous leprosy in treatment
* age between 20 and 60
* body mass index (BMI) between 18 and 35 kg/m2
* ability to follow given directions and to attend assessments and
* Fitzpatrick's Phototype I-IV

Exclusion Criteria:

* females
* arterial hypertension
* diabetes mellitus
* BMI greater than 35 kg/m2
* collagenosis
* past or present history of smoking
* age under 20 and over 60 years.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2006-03; Primary Completion 2009-11 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Laser-Doppler flowmetry | 0 - 20 min.
  perfusion units (PU: 1 PU=10 mV)

SECONDARY OUTCOMES:
Cytoscan | 0 - 5min
  Using the Cystoscan, we have evaluated functional capillary density, diameter of the dermal papilla, capillary diameter, capillary handle diameter and capillary morphology

CONTACTS AND LOCATIONS:
Overall Officials: curt treu, PhD, Principal Investigator — Rio de Janeiro State University; Eliete Bouskela, PhD, Study Director — Rio de Janeiro State University